CLINICAL TRIAL: NCT04596436
Title: Patterns of Injury and Mortality in Free-fall Trauma Patients: a Multi-center Study
Brief Title: Mortality in Free-fall Trauma Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202009091RINC
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2021-11

CONDITIONS: Free Fall Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
In this study, the investigators aimed to analyze the demographic characteristics, patterns of injury, and mortality after free fall in the emergency department of the National Taiwan University Hospital, and the affiliations, Hsin-Chu branch, and Yun-lin branch.

DETAILED DESCRIPTION:
Falls from a height are the leading cause of accidental deaths. The mechanism of free-fall injury is abrupt vertical deceleration and the severity is dependent on the height, body weight, posture and contact area…etc. Most victims presented to the emergency department with major trauma, so initial evaluation and management are crucial for survival. The knowledge of the unique pattern of injuries helps clinicians to facilitate the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

patients aged more than 20 years after free falls in the emergency department of the National Taiwan University Hospital, and the affiliations, Hsin-Chu branch, and Yun-lin branch.

Exclusion Criteria:

patients aged less than 20 years after free fall in the emergency department of the National Taiwan University Hospital, and the affiliations, Hsin-Chu branch, and Yun-lin branch.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged more than 20 years after free falls in the emergency department of the National Taiwan University Hospital, and the affiliations, Hsin-Chu branch, and Yun-lin branch.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
mortality after free falls | 60 days
  death rate

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — NTUH
Locations (1):
- Wan-Ching Lien, Taipei, Taiwan